CLINICAL TRIAL: NCT05636852
Title: An Open-label Multicenter Phase 2 Dose-evaluation Study of Altropane (123I) Injection for Striatal Dopamine Transporter Visualization Using SPECT Brain Imaging
Brief Title: Altropane Dose for Imaging Patients With Suspected Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: GE Healthcare (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-278-001
Record Dates: First submitted 2022-11-01; First posted 2022-12-05 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: SPECT; Altropane; Parkinson's disease; Parkinsonian syndromes; movement disorders; striatum; dopamine transporter
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Parkinsonian Disorders | interventions — N-iodoallyl-2-carbomethoxy-3-(4-fluorophenyl)tropane; Iodine-123; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Altropane (123I) Injection (Experimental)
  Interventions: Drug: Altropane (123I) Injection

INTERVENTIONS:
Drug: Altropane (123I) Injection — Each participant received a single intravenous (IV) administration of 5 millicuries (mCi) (185 megabecquerels [MBq]) of Altropane (123I) Injection on Day 1. Altropane SPECT images were acquired for 30 minutes starting 15 to 20 minutes after administration with Altropane. These images were visually interpreted by 5 expert independent blinded readers.

SUMMARY:
Previous studies showed that a dose of 8 millicuries of Altropane was appropriate for imaging patients with suspected Parkinson's disease. This study determined if a lower dose (5 millicuries) would suffice.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1: a) the participant had a DaTscan image, obtained within 1 year (preferably within 6 months) before screening, that showed normal striatal uptake and b) the participant had a clinical diagnosis (made by a board-certified neurologist who was qualified by training and experience in the diagnosis of movement disorders) that was consistent with the DaTscan image.

For Part 2 (which was not conducted): a) the participant had a DaTscan image, obtained within 1 year (preferably within 6 months) before screening, that showed abnormal (unilateral or bilateral reduced) striatal uptake and b) the participant also had a confirmed clinical diagnosis of a dPS (such as Parkinson's disease, multiple system atrophy, corticobasal degeneration, progressive supranuclear palsy, etc.) made by a board-certified neurologist who was qualified by training and experience in the diagnosis of movement disorders, and c) the diagnosis was consistent with the DaTscan image.

* The participant was male or female, ≥18 years of age, of any race and ethnicity.
* The participant was able and willing to comply with study procedures and signed and dated informed consent was obtained.
* If the participant was a woman of childbearing potential*, she must have used a highly effective method of contraception** from Screening until 30 days after the last administration of Altropane, and the results of a serum or urine human chorionic gonadotropin (hCG) pregnancy test, performed at Screening and on the day of Altropane administration (with the result known before Altropane administration), must have been negative.

  * A woman of childbearing potential was defined as neither post-menopausal nor surgically sterile. Post-menopausal means having had no menses for at least 12 months without an alternative medical cause. Surgically sterile means having had a documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, or any combination of these.

  ** A highly effective method of contraception was defined as one that had a failure rate of less than 1% per year when used consistently and correctly; such methods included combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable); intrauterine device; intrauterine hormone-releasing system; bilateral tubal ligation/occlusion; vasectomized partner (with medical confirmation of success); and abstinence from heterosexual intercourse involving a woman of childbearing potential.
* If the participant was a male*** with a sexual partner who was a woman of childbearing potential*, he and his partner must have used adequate contraception** from Screening until 30 days after the last administration of Altropane.

(***A male was considered fertile after puberty unless permanently sterile by bilateral orchidectomy, or vasectomized with confirmation of success.)

Exclusion Criteria:

* The participant was previously included in this study.
* Fewer than 7 disintegration half-lives had elapsed between the participant's last procedure (therapeutic or diagnostic) involving a radioisotope and Visit 2 (altropane SPECT imaging).
* Including participation in this study, the participant's total exposure to radiation during medical procedures/tests in the past year would have exceeded 50 mSv.
* The participant had participated in an investigational drug or device clinical trial within 30 days before the date of informed consent.
* The participant had any clinically significant or unstable physical or psychological illness, structural brain abnormality, abnormal laboratory results, or abnormal ECG (based on medical history or physical examination at Screening), as determined by the Principal Investigator, that would interfere with study participation.
* The participant had any history of drug or alcohol abuse in the 2 years prior to the date of informed consent.
* The participant had a positive urine screen for drugs of abuse at Screening.
* The participant was a pregnant or breast-feeding female, or was a female of child-bearing potential that was not using appropriate birth control.
* The participant was unable to lie supine for 1 hour.
* The participant had any thyroid disease other than adequately treated hypothyroidism.
* The participant had known or suspected allergy/hypersensitivity to any ingredient in Altropane or to the thyroid blocking medication to be used before imaging.
* The participant was taking any of the medications/treatments listed in the protocol as disallowed and could not or would not discontinue use at least 12 hours prior to SPECT exam.
* The participant was referred to DaTscan imaging for evaluation of possible cognitive impairment including dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, MD, PhD, Study Director — GE Healthcare
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 24 April 2023 to 08 June 2024 at 4 centers in the United States.
Pre-assignment Details: A total of 15 eligible participants entered in Part 1 of study. 13 participants received a single dose of Altropane. Two subjects were not dosed due to scheduling issues. The study was planned to be conducted in 2 parts. However, due to business decisions the sponsor terminated the study after completion of Part 1. This decision was not due to safety concerns.
Groups:
- Part 1: Altropane (123I) Injection: Each participant received a single intravenous (IV) administration of 5 millicuries (mCi) (185 megabecquerels [MBq]) of Altropane (123I) Injection on Day 1. Altropane SPECT images were acquired for 30 minutes starting 15 to 20 minutes after administration with Altropane. These images were visually interpreted by 5 independent expert blinded readers.
Period: Overall Study
Arm/Group | Part 1: Altropane (123I) Injection
Started | 15
Safety Set (Safety Analysis Set consisted of all participants who received a single dose of Altropane.) | 13
Full Analysis Set (Full Analysis Set consisted of all participants who received any amount of Altropane and had an Altropane image interpretation.) | 10
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other than specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Striatal Visualization: Percentage of Participants With Correct Majority Classifications of 5-mCi Altropane Images as Determined by 5 Independent Blinded Readers
Description: Assessment of the Altropane SPECT images was performed by 5 independent expert blinded readers to determine striatal uptake, reported as a forced choice of either normal (caudate and putamen fully visible on left and right, or with small insignificant defects) or abnormal (unilateral or bilateral reduced). Majority classification was determined from the majority interpretation of the 5 expert blinded readers (at least 3 of 5 readers).
Time Frame: Day 1, up to 30 minutes
Population: Full Analysis Set consisted of all participants who received any amount of Altropane and had an Altropane image interpretation.
Measure: Number; unit: percentage of participants
Groups:
- Part 1: Altropane (123I) Injection: Each participant received a single intravenous (IV) administration of 5 millicuries (mCi) (185 megabecquerels [MBq]) of Altropane (123I) Injection on Day 1. Altropane SPECT images were acquired for 30 minutes starting 15 to 20 minutes after administration with Altropane. These images were visually interpreted by 5 expert independent blinded readers.
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 10
percentage of participants
  Reader 1 | 60
  Reader 2 | 80
  Reader 3 | 90
  Reader 4 | 70
  Reader 5 | 80
  Majority Readers | 80

2. Secondary Outcome: Percentage of Participants With Confidence Ratings for 5-mCi Altropane Images as Evaluated by 5 Independent Blinded Readers (Reader Confidence in Striatal Visualization)
Description: Visual interpretation of the Altropane SPECT images was conducted by 5 independent expert readers who were blinded to each participant's clinical information, and who were not otherwise involved in the study. Their visual image interpretations were a forced choice between normal (caudate and putamen fully visible on left and right, or with small insignificant defects) or abnormal (unilateral or bilateral reduced) striatal uptake. Readers evaluated their confidence in striatal visualization, rating it as high, medium, or low. Majority classification was determined from the majority interpretation of the 5 expert blinded readers (at least 3 of 5 readers) using the high and medium/low groupings. Percentage of participants with confidence ratings for 5-mCi Altropane images are reported.
Time Frame: Day 1, up to 30 minutes
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 10
percentage of participants
  Reader 1 : High | 40
  Reader 1 : Medium | 40
  Reader 1 : Low | 20
  Reader 2 : High | 80
  Reader 2 : Medium | 20
  Reader 2 : Low | 0
  Reader 3 : High | 70
  Reader 3 : Medium | 30
  Reader 3 : Low | 0
  Reader 4 : High | 90
  Reader 4 : Medium | 10
  Reader 4 : Low | 0
  Reader 5 : High | 50
  Reader 5 : Medium | 40
  Reader 5 : Low | 10

3. Secondary Outcome: Percentage of Participants With Image Quality for 5-mCi Altropane Images as Evaluated by 5 Independent Blinded Readers (Reader Assessment of Image Quality)
Description: Visual interpretation of the Altropane SPECT images was conducted by 5 independent expert readers who were blinded to each participant's clinical information, and who were not otherwise involved in the study. Their visual image interpretations were a forced choice between normal (caudate and putamen fully visible on left and right, or with small insignificant defects) or abnormal (unilateral or bilateral reduced) striatal uptake. Readers assessed image quality as excellent, good, fair, poor, or unevaluable. Majority classification was determined from the majority interpretation of the 5 expert blinded readers (at least 3 of 5 readers) using the excellent/good and fair/poor/unevaluable groupings. Percentage of participants with image quality for 5-mCi Altropane images are reported.
Time Frame: Day 1, up to 30 minutes
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 10
percentage of participants
  Reader 1 : Excellent | 90
  Reader 1 : Good | 0
  Reader 1 : Fair | 10
  Reader 1 : Unevaluable | 0
  Reader 2 : Excellent | 70
  Reader 2 : Good | 30
  Reader 2 : Fair | 0
  Reader 2 : Unevaluable | 0
  Reader 3 : Excellent | 80
  Reader 3 : Good | 20
  Reader 3 : Fair | 0
  Reader 3 : Unevaluable | 0
  Reader 4 : Excellent | 60
  Reader 4 : Good | 40
  Reader 4 : Fair | 0
  Reader 4 : Unevaluable | 0
  Reader 5 : Excellent | 20
  Reader 5 : Good | 50
  Reader 5 : Fair | 30
  Reader 5 : Unevaluable | 0

4. Secondary Outcome: Inter-Reader Agreement on Percentage of Participants With Normal Images
Description: Visual interpretation of the Altropane SPECT images was conducted by 5 independent expert readers who were blinded to each subject's clinical information, and who were not otherwise involved in the study. Their visual image interpretations were a forced choice between normal (caudate and putamen fully visible on left and right, or with small insignificant defects) or abnormal (unilateral or bilateral reduced) striatal uptake. Percentage of participants with inter-reader agreement on striatal visualization classification for whom 5, 4, and 3 readers, respectively, were in agreement on the participants classification (normal images) are reported.
Time Frame: Day 1, up to 30 minutes
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 10
percentage of participants
  5 Readers in Agreement | 70
  4 Readers in Agreement | 20
  3 Readers in Agreement | 10

5. Secondary Outcome: Percentage of Participants With One or More Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product, which did not necessarily have a causal relationship with the treatment. Treatment-Emergent Adverse Events (TEAEs) were defined as AEs that started or worsened between the start of pharmaceutical product administration and the end of the follow-up period.
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
percentage of participants | 23.1

6. Secondary Outcome: Percentage of Participants With Adverse Drug Reaction (ADR)
Description: ADR is an AE that is caused by the investigational medicinal product.
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
percentage of participants | 0

7. Secondary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Percentage of participants with clinically significant changes from baseline in vital signs (systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature). Normal limits of vital signs are:
  1. Systolic BP (mmHg) - low: 85 and High: 139; Diastolic BP (mmHg) - low: 60 and High: 89.
  2. Heart rate (bpm) - low: 60 and High: 100.
  3. Respiration Rate (rpm) - low: 12 and High: 22.
  4. Body Temperature - low: 36.4 degree Celsius (97.5 degree Fahrenheit) and High: 37.7 degree Celsius (99.5 degree Fahrenheit).
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
percentage of participants | 0

8. Secondary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Physical Examination Until 24 Hours Post Dose
Description: Percentage of participants with clinically significant changes from baseline in physical examination (general appearance, lungs and heart).
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
Percentage of participants | 0

9. Secondary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Electrocardiogram (ECG) Examinations (PR Interval, QTc, QRS and RR Interval) Until 24 Hours Post Dose
Description: Percentage of participants with clinically significant changes from baseline in electrocardiogram (ECG) examinations: (PR interval, QTc, QRS and RR interval). The normal limits (ms) of ECG variables:
  1. PR interval (ms) - low: 120 and high: 200
  2. QRS interval (ms) - low: 50 and high: 100
  3. QTc interval (ms)- high =<440
  4. RR interval (ms) - low: 600 and high: 1000
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
percentage of participants | 0

10. Secondary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Serum Biochemistry and Hematology Parameters Until 24 Hours Post Dose
Description: Percentage of participants with clinically significant changes from baseline in serum biochemistry (Alanine aminotransferase, Albumin, Alkaline phosphatase, Bicarbonate, Creatine phosphokinase (CPK), total Creatinine, Protein (total), Phosphorous Glucose) and hematology parameters (Red blood cell (RBC) count, Platelet count, White blood cell (WBC) count).
Time Frame: From administration of Altropane until 24 hours post dose
Population: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Altropane (123I) Injection
Number analyzed (Participants) | 13
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: From administration of Altropane until 24 hours post dose
Description: Safety Analysis Set consisted of all participants who received a single dose of Altropane.
Arm/Group | Part 1: Altropane (123I) Injection
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Altropane (123I) Injection (N=13)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated after completion of Part 1 by the Sponsor due to business decision. This decision was not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT05636852/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT05636852/SAP_001.pdf